CLINICAL TRIAL: NCT04793945
Title: The Efficacy of Combining 308 Nm-Excimer Light and Topical Steroid in the Treatment of Alopecia Areata
Brief Title: Excimer Light and Topical Steroid in Treatment of Alopecia Areata
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, fatma magdy zidan taraaf, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fmztaraaf
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: patients with three patches of Alopecia Areata the first patch will be treated by topical steroid and Excimer light the second patch will be treated by topical steroid only the third patch will be left as a control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light therapy twice weekly (Active Comparator): 15 or half of the patients with three patches of Alopecia Areata on the scalp the first patch will be treated by 308nm Excimer light twice weekly and topical steroid twice daily the second patch will be treated by topical steroid twice daily. the third patch will be left as a control.
  Interventions: Combination Product: topical steroid and 308nm-Excimer light therapy
- light therapy once weekly (Active Comparator): 15 or half of the patients with three patches of Alopecia Areata on the scalp the first patch will be treated by 308nm Excimer light once weekly and topical steroid twice daily.
  the second patch will be treated by topical steroid twice daily. the third patch will be left as a control.
  Interventions: Combination Product: topical steroid and 308nm-Excimer light therapy

INTERVENTIONS:
Combination Product: topical steroid and 308nm-Excimer light therapy — applying topical steroid in combination with 308nm-Excimer light therapy to treat Alopecia Areata

SUMMARY:
Alopecia areata is a polygenic autoimmune disease causing hair loss, particularly during the anagen phase of hair growth This condition has a lifetime risk of about 2.1% of the world population and the cumulative incidence seems to rise linearly with age .

Patchy non scarring hair loss on the scalp is the most common clinical presentation, although it can also occur elsewhere . In addition to patchy Alopecia Areata , a more severe form, alopecia totalis , presents with diffuse hair loss across the scalp. In the most severe form, alopecia universalis , hair loss occurs on all areas of the body, including the beard, eyelashes, and extremities .

DETAILED DESCRIPTION:
Alopecia Areata can have a large impact on patients' quality of life, causing both cosmetic and psychosocial distress. Studies on the impact of hair loss have shown high levels of self-consciousness, jealousy, embarrassment, depression, introversion, and decreased self-esteem .

Alopecia Areata can occur at any age, but it is most common among young and middle-aged people . Both sexes are equally affected. Several environmental factors have been suggested as triggering Alopecia Areata, including infection, drugs, trauma, and stress. Thyroid autoimmune disease, atopy, and vitiligo are commonly associated. Diverse physical or psychological insults may trigger the episodes of Alopecia Areata, but there is no evidence that they influence prognosis.

Etiology of Alopecia Areata is not completely understood, and the majority of evidence suggests that genetically predisposed individuals, when exposed to an unknown trigger, develop a predominantly autoimmune reaction, leading to acute hair loss.

Although many patients improve spontaneously or respond to standard therapy, treatment can be quite challenging in those with more severe and refractory disease .

Topical corticosteroids are often the first line of treatment for mild patchy alopecia, with the underlying mechanism being containment of inflammation and hastening of the recovery of damaged hair follicles . Additionally, corticosteroids may be delivered via intralesional injection with slightly better effects (63% with complete regrowth within 4 months in one study . However, this method cannot be used for rapidly progressing variants and does not prevent hair loss at other sites . Furthermore, both topical and intralesional steroids increase the risk of cutaneous atrophy at the site of treatment, and intralesional steroids may decrease bone mineral density .

With the development of new technologies, more and more lasers or lamps have been used to treat alopecia, such as ultraviolet , Excimer laser/lamp , low-level laser , erbium-glass laser, thulium laser , and carbon dioxide laser . Individual researchers have been considering 308-nm Excimer lamp to be used for treating Alopecia Areata by inducing apoptosis of T lymphocytes, but the effective rates had differences in studies .

Excimer laser using high-dose monochromatic UV radiation can trigger apoptosis and induce immunological suppression through altering cytokine production such as interleukin-4, interleukin-10, prostaglandin E2, platelet-activating factor, and cis-urocanic acid .

ELIGIBILITY:
Inclusion Criteria:

* aged 16-40 years,
* Good general health,
* A clinical diagnosis of multiple Alopecia Areata of the scalp.
* Hair loss <25 percent of the total scalp.
* No use of drugs or hair care products influencing hair growth in the last 2 months.

Exclusion Criteria:

* Other causes of hair loss (like endocrine or immunological diseases).
* Skin disease in the treatment area.
* Pregnant or lactating patients.
* Hair transplantation history.
* Photosensitivity history.
* Malignant tumor history.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Severity of ALopecia Tool score | 9months
  The scalp is divided into four parts on the basis of surface area as follows: vertex or top = 40 percent (0.40), right side = 18 percent (0.18), left side = 18 percent (0.18) and the posterior aspect = 24 percent (0.24). Percentage of hair loss in any of the four areas was multiplied by the percentage of the scalp covered in that area. The Severity of Alopecia Tool score is the sum of the percentage of hair loss in all the areas mentioned above.[10]
digital photographs | 9months
  using identical camera settings, lighting, patient positioning and background.
The hair regrowth in the patches of alopecia | 9months
  0 = no hair regrowth,
  1. = 1-25percent hair regrowth,
  2. = 26-50percent hair regrowth,
  3. = 51-75percent hair regrowth, and
  4. = 76-100 percent hair regrowth.
Dermoscopic evaluation | 9months
  Dermoscopy will be used to analyze the change in the count of hair at intervals of 4 weeks. The number of hair (total, vellus, and terminal hairs) will be calculated by dermoscopy .
A patient satisfaction score | 9months
  0 to 25percent change = not satisfied, 26 to 50percent = mildly satisfied, 51 to 75percent = moderately satisfied, 76 to 100percent = very satisfied
adverse effects | 9months
  Any encountered adverse effects in terms of pain, erythema, edema and crusts will be recorded.
dermoscopic evaluation | 9months
  The mean diameter of hair will be recorded for analysis.
dermoscopic evaluation | 9months
  diameter of hair will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Fatma m zidan, student, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: one year

REFERENCES:
- [Background] Pratt CH, King LE Jr, Messenger AG, Christiano AM, Sundberg JP. Alopecia areata. Nat Rev Dis Primers. 2017 Mar 16;3:17011. doi: 10.1038/nrdp.2017.11. PMID 28300084
- [Background] Mirzoyev SA, Schrum AG, Davis MDP, Torgerson RR. Lifetime incidence risk of alopecia areata estimated at 2.1% by Rochester Epidemiology Project, 1990-2009. J Invest Dermatol. 2014 Apr;134(4):1141-1142. doi: 10.1038/jid.2013.464. Epub 2013 Nov 11. No abstract available. PMID 24202232
- [Background] Villasante Fricke AC, Miteva M. Epidemiology and burden of alopecia areata: a systematic review. Clin Cosmet Investig Dermatol. 2015 Jul 24;8:397-403. doi: 10.2147/CCID.S53985. eCollection 2015. PMID 26244028
- [Background] Hordinsky MK. Overview of alopecia areata. J Investig Dermatol Symp Proc. 2013 Dec;16(1):S13-5. doi: 10.1038/jidsymp.2013.4. PMID 24326541
- [Background] Girman CJ, Hartmaier S, Roberts J, Bergfeld W, Waldstreicher J. Patient-perceived importance of negative effects of androgenetic alopecia in women. J Womens Health Gend Based Med. 1999 Oct;8(8):1091-5. doi: 10.1089/jwh.1.1999.8.1091. PMID 10565667
- [Background] Wells PA, Willmoth T, Russell RJ. Does fortune favour the bald? Psychological correlates of hair loss in males. Br J Psychol. 1995 Aug;86 ( Pt 3):337-44. doi: 10.1111/j.2044-8295.1995.tb02756.x. PMID 7551645
- [Background] Al Hamzawi NK. Evaluation of the Efficacy and Safety of 308-nm Monochromatic Excimer Lamp in the Treatment of Resistant Alopecia Areata. Int J Trichology. 2019 Sep-Oct;11(5):199-206. doi: 10.4103/ijt.ijt_74_19. PMID 31728102
- [Background] McElwee KJ, Gilhar A, Tobin DJ, Ramot Y, Sundberg JP, Nakamura M, Bertolini M, Inui S, Tokura Y, King LE Jr, Duque-Estrada B, Tosti A, Keren A, Itami S, Shoenfeld Y, Zlotogorski A, Paus R. What causes alopecia areata? Exp Dermatol. 2013 Sep;22(9):609-26. doi: 10.1111/exd.12209. PMID 23947678
- [Background] Olsen EA, Hordinsky MK, Price VH, Roberts JL, Shapiro J, Canfield D, Duvic M, King LE Jr, McMichael AJ, Randall VA, Turner ML, Sperling L, Whiting DA, Norris D; National Alopecia Areata Foundation. Alopecia areata investigational assessment guidelines--Part II. National Alopecia Areata Foundation. J Am Acad Dermatol. 2004 Sep;51(3):440-7. doi: 10.1016/j.jaad.2003.09.032. No abstract available. PMID 15337988
- [Background] Messenger AG, McKillop J, Farrant P, McDonagh AJ, Sladden M. British Association of Dermatologists' guidelines for the management of alopecia areata 2012. Br J Dermatol. 2012 May;166(5):916-26. doi: 10.1111/j.1365-2133.2012.10955.x. No abstract available. PMID 22524397
- [Background] 12. Kranseler, J. S. & Sidbury, R. 2017. Alopecia Areata: Update on Management. Indian Journal of Paediatric Dermatology, 18, 261.
- [Background] Charuwichitratana S, Wattanakrai P, Tanrattanakorn S. Randomized double-blind placebo-controlled trial in the treatment of alopecia areata with 0.25% desoximetasone cream. Arch Dermatol. 2000 Oct;136(10):1276-7. doi: 10.1001/archderm.136.10.1276. No abstract available. PMID 11030789
- [Background] Kubeyinje EP. Intralesional triamcinolone acetonide in alopecia areata amongst 62 Saudi Arabs. East Afr Med J. 1994 Oct;71(10):674-5. PMID 7821250
- [Background] Samrao A, Fu JM, Harris ST, Price VH. Bone mineral density in patients with alopecia areata treated with long-term intralesional corticosteroids. J Drugs Dermatol. 2013 Feb;12(2):e36-40. PMID 23377403
- [Background] Herz-Ruelas ME, Welsh O, Gomez-Flores M, Welsh E, Miranda-Maldonado I, Ocampo-Candiani J. Ultraviolet A-1 phototherapy as an alternative for resistant alopecia areata. Int J Dermatol. 2015 Oct;54(10):e445-7. doi: 10.1111/ijd.13054. No abstract available. PMID 26394604
- [Background] El Taieb MA, Hegazy EM, Ibrahim HM, Osman AB, Abualhamd M. Topical calcipotriol vs narrowband ultraviolet B in treatment of alopecia areata: a randomized-controlled trial. Arch Dermatol Res. 2019 Oct;311(8):629-636. doi: 10.1007/s00403-019-01943-8. Epub 2019 Jun 24. PMID 31236672
- [Background] Darwin E, Arora H, Hirt PA, Wikramanayake TC, Jimenez JJ. A review of monochromatic light devices for the treatment of alopecia areata. Lasers Med Sci. 2018 Feb;33(2):435-444. doi: 10.1007/s10103-017-2412-6. Epub 2017 Dec 17. PMID 29250710
- [Background] Panchaprateep R, Pisitkun T, Kalpongnukul N. Quantitative proteomic analysis of dermal papilla from male androgenetic alopecia comparing before and after treatment with low-level laser therapy. Lasers Surg Med. 2019 Sep;51(7):600-608. doi: 10.1002/lsm.23074. Epub 2019 Mar 7. PMID 30843235
- [Background] Esmat SM, Hegazy RA, Gawdat HI, Abdel Hay RM, Allam RS, El Naggar R, Moneib H. Low level light-minoxidil 5% combination versus either therapeutic modality alone in management of female patterned hair loss: A randomized controlled study. Lasers Surg Med. 2017 Nov;49(9):835-843. doi: 10.1002/lsm.22684. Epub 2017 May 10. PMID 28489273
- [Background] Al-Dhalimi MA, Al-Janabi MH, Abd Al Hussein RA. The Use of a 1,540 nm Fractional Erbium-Glass Laser in Treatment of Alopecia Areata. Lasers Surg Med. 2019 Dec;51(10):859-865. doi: 10.1002/lsm.23133. Epub 2019 Jul 18. PMID 31321800
- [Background] Cho SB, Goo BL, Zheng Z, Yoo KH, Kang JS, Kim H. Therapeutic efficacy and safety of a 1927-nm fractionated thulium laser on pattern hair loss: an evaluator-blinded, split-scalp study. Lasers Med Sci. 2018 May;33(4):851-859. doi: 10.1007/s10103-018-2437-5. Epub 2018 Jan 16. PMID 29340854
- [Background] Majid I, Jeelani S, Imran S. Fractional Carbon Dioxide Laser in Combination with Topical Corticosteroid Application in Resistant Alopecia Areata: A Case Series. J Cutan Aesthet Surg. 2018 Oct-Dec;11(4):217-221. doi: 10.4103/JCAS.JCAS_96_18. PMID 30886476
- [Background] McMichael AJ. Excimer laser: a module of the alopecia areata common protocol. J Investig Dermatol Symp Proc. 2013 Dec;16(1):S77-9. doi: 10.1038/jidsymp.2013.31. PMID 24326569
- [Background] Li A, Meng X, Xing X, Tan H, Liu J, Li C. Efficacy and Influence Factors of 308-nm Excimer Lamp with Minoxidil in the Treatment of Alopecia Areata. Lasers Surg Med. 2020 Oct;52(8):761-767. doi: 10.1002/lsm.23210. Epub 2020 Jan 9. PMID 31919885